CLINICAL TRIAL: NCT01557361
Title: STandard Versus Accelerated Initiation of Renal Replacement Therapy in Acute Kidney Injury (STARRT-AKI)
Brief Title: Standard Versus Accelerated Initiation of Dialysis in Acute Kidney Injury
Acronym: STARRT-AKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alere San Diego (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR MOP 111116
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2013-08

CONDITIONS: Acute Kidney Injury
Keywords: renal replacement therapy; dialysis; acute kidney injury; hemodialysis; critical illness
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard RRT initiation (Active Comparator): RRT is initiated >12 hours after eligibility determination. Once a decision is made to start RRT, a dialysis catheter will be placed and RRT initiated as soon as possible.
  Interventions: Other: Standard RRT initiation
- Accelerated RRT initiation (Experimental): A dialysis catheter will be placed and RRT initiated as soon as possible and within 12 hours of eligibility.
  Interventions: Other: Accelerated RRT initiation

INTERVENTIONS:
Other: Accelerated RRT initiation — A dialysis catheter will be placed and RRT initiated as soon as possible and within 12 hours of eligibility. This 12 hour window includes the time needed to obtain consent.
  Arms: Accelerated RRT initiation
Other: Standard RRT initiation — Patients will be carefully followed over a period of 7 days to identify potential indications for RRT. The trial team will ask that the clinical team consider RRT initiation if there are:
  I. Criteria for persistent AKI (serum creatinine has not declined by more than 50% from value recorded at time of eligibility) AND
  II. At least one of the following indications for RRT initiation:
  1. Serum potassium ≥6.0 mmol/L, or
  2. Serum bicarbonate ≤ 10 mmol/L, or
  3. Evidence of severe respiratory failure, based on a PaO2/FiO2 <200 and bilateral infiltrates on the chest x-ray, or
  4. By 72 hours after randomization, creatinine has not declined by more than 50% from that recorded at the time of randomization
  Arms: Standard RRT initiation

SUMMARY:
The objectives of this trial are to determine whether, in critically ill patients with severe acute kidney injury (AKI), randomization to accelerated initiation of renal replacement therapy (RRT), compared with standard initiation, is:

1. Feasible, in terms of adherence to the protocol (primary outcome), recruitment rates, and achievement of follow-up; and
2. Safe, from the perspective of potential adverse events associated with earlier initiation of RRT

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common and devastating complication of critical illness. Once AKI is established, treatment is largely supportive and no intervention has been found to restore kidney function or improve overall survival. Renal replacement therapy (RRT), usually in the form of hemodialysis, is frequently needed to manage patients with severe AKI. Such patients have an in-hospital mortality that consistently exceeds 50%. Delay in the initiation of RRT has been implicated as a possible contributor to this poor outcome. A recent meta-analysis suggested that earlier initiation of RRT may improve survival. However, completed trials to date have been small, single centre, limited by study quality, and have shown considerable heterogeneity in terms of definitions used for "early" RRT initiation.

The objectives of this trial are to determine whether, in critically ill patients with severe acute kidney injury (AKI), randomization to accelerated initiation of renal replacement therapy (RRT), compared with standard initiation, is:

1. Feasible, in terms of adherence to the protocol (primary outcome), recruitment rates, and achievement of follow-up; and
2. Safe, from the perspective of potential adverse events associated with the earlier or later initiation of RRT

This pilot trial is intended to guide and inform the design of a phase III multicentre randomized trial of accelerated versus standard initiation of RRT in critically ill patients that will evaluate the impact of the intervention on 90-day all-cause mortality and recovery of kidney function.

ELIGIBILITY:
Inclusion Criteria (all of these need to be present):

1. Age ≥ 18 years
2. Admission to an intensive care unit
3. Evidence of kidney dysfunction (serum creatinine ≥ 100 µmol/L (women) or

   ≥ 130 µmol/L (men))
4. Evidence of severe AKI defined by at least 2 of the following 3 criteria:

   i-A 2-fold increase in serum creatinine during hospitalization or from a known pre-hospitalization baseline ii-Oliguria as defined by total urine output < 6 mL/kg over the preceding 12 hours iii-Whole blood Neutrophil Gelatinase-Associated Lipocalin (NGAL) ≥ 400ng/mL
5. Likelihood that an absolute indication for RRT will not arise in the subsequent 24 hours based on the most recent bloodwork for the following parameters: i- Serum potassium ≤ 5.5 mmol/L and ii- Serum bicarbonate ≥ 15 mmol/L
6. Central venous pressure ≥ 8 mmHg

Exclusion Criteria (the presence of one of these would disqualify eligibility):

1. Lack of commitment to ongoing life support
2. Presence of a drug overdose that necessitates initiation of RRT
3. Any RRT within the previous 2 months
4. Presence or clinical suspicion of renal obstruction, rapidly progressive glomerulonephritis, vasculitis, or acute interstitial nephritis
5. Advanced chronic kidney disease, defined by an estimated glomerular filtration rate < 30 mL/min/1.73 m2, based on pre-hospitalization blood work
6. Kidney transplant within the past 365 days
7. At the time of screening, doubling of serum creatinine has been present for > 48 hours
8. Clinician(s) caring for patient believe(s) that immediate dialysis is absolutely mandated
9. Clinician(s) caring for patient believe(s) that deferral of dialysis initiation is mandated
10. Patient or substitute decision maker can not provide consent within 12 hours of study eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of protocol adherence | 14 days
  >90% of participants in the accelerated initiation arm start RRT within 12 hours of eligibility AND >90% of participants randomized to the standard initiation arm who ultimately receive RRT, start RRT at least 12 hours following eligibility determination

SECONDARY OUTCOMES:
Feasibility of enrollment | 14 days
  >50% of eligible patients are successfully enrolled in the trial
Feasibility of 90-day follow-up | 90 days
  Vital status and need for RRT at 90 days are successfully captured in >95% of participants
Safety outcomes | 14 days
  Serious adverse effects, with a particular focus on those that are potentially attributable to the study treatment, vascular accesss complications (including hemorrhage, thrombosis and infection) and complications associated with the delivery of RRT (dialysis-associated hypotension, electrolyte abnormalities) will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wald, MDCM MPH, Principal Investigator — Unity Health Toronto; Sean M Bagshaw, MD MSc, Principal Investigator — University of Alberta
Locations (11):
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre hopitalier universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Wing S, Neto AS, Bellomo R, Clark EG, Gallagher M, Liangos O, Prasad B, Silver SA, Tolwani A, Bagshaw S, Wald R. CKD Progression after Acute Kidney Injury: A Secondary Analysis of the Standard versus Accelerated Initiation of Renal Replacement Therapy in Acute Kidney Injury Trial. Kidney360. 2025 Apr 1;6(4):636-644. doi: 10.34067/KID.0000000663. Epub 2024 Dec 3. PMID 39625781
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Smith OM, Wald R, Adhikari NK, Pope K, Weir MA, Bagshaw SM; Canadian Critical Care Trials Group. Standard versus accelerated initiation of renal replacement therapy in acute kidney injury (STARRT-AKI): study protocol for a randomized controlled trial. Trials. 2013 Oct 5;14:320. doi: 10.1186/1745-6215-14-320. PMID 24093950